CLINICAL TRIAL: NCT02310321
Title: A Phase 1/2 Study of ASP2215 in Combination With Induction and Consolidation Chemotherapy in Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: A Study of ASP2215 in Combination With Induction and Consolidation Chemotherapy in Patients With Newly Diagnosed Acute Myeloid Leukemia.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-0104
Record Dates: First submitted 2014-12-01; First posted 2014-12-08 (Estimated); Results first posted 2024-10-16 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia; FLT3-mutated Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Cytarabine; Idarubicin; ASP2215
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib; Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Phase 1: Dose Evaluation (DEv) (Experimental): Induction period: Participants received 120 milligrams (mg) gilteritinib (3 tablets of 40 mg) orally, once daily from day 4 to 17 combined with chemotherapy (idarubicin: 12 mg per square meters per day [mg/m^2/day] on days 1 to 3, cytarabine: 100 mg/m^2/day on days 1 to 7) via intravenous (IV) infusion; in cycles (C) 1 and 2 (1 cycle= 42 days).
  Consolidation period: Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once daily from day 1 to 14 combined with chemotherapy (cytarabine: 1500 mg/m^2, twice daily on days 1, 3, and 5) via IV infusion; in the consolidation period in C1 to 3 (1 cycle= 28 days).
  Duration of infusion was determined by site clinical practice and local package insert in both induction and consolidation periods..
  Maintenance period: Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once daily from days 1 to 28 in the maintenance period in C1 to 26 or untill discontinuation criterion is met (1 cycle= 28 days).
  Interventions: Drug: Gilteritinib; Drug: Idarubicin; Drug: Cytarabine
- Phase 1: Dose Expansion (DEx) (Experimental): Induction period: Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 4 to 17 in combination with chemotherapy (idarubicin: 12 mg/m^2/day on days 1 to 3, cytarabine: 100 mg/m^2/day on days 1 to 7) via IV infusion; in the induction period in C1 and 2 (1 cycle= 42 days).
  Consolidation period: Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 1 to 14 in combination with chemotherapy (cytarabine: 1500 mg/m^2, twice daily on days 1, 3, and 5) via IV infusion; in the consolidation period in C1 to 3 (1 cycle= 28 days).
  Duration of infusion was determined based on site clinical practice and the local package insert in both induction and consolidation periods.
  Maintenance period: Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 1 to 28 in the maintenance period in C1 to 26 or a discontinuation criterion is met (1 cycle= 28 days).
  Interventions: Drug: Gilteritinib; Drug: Idarubicin; Drug: Cytarabine
- Phase 2: FLT3-mutated AML (Experimental): Induction period: Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once daily from days 8 until blood recovery combined with chemotherapy (idarubicin: 12 mg/m^2/day on days 1 to 3, cytarabine: 100 mg/m^2/day on days 1 to 7) via IV infusion; in C1 and 2. Each cycle was extended until blood recovery was observed.
  Consolidation period: Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once daily from days 1 until blood recovery combined with chemotherapy (cytarabine: 1500 mg/m^2, twice daily on days 1, 3, and 5) via IV infusion; in C1 to 3. Each cycle was extended until blood recovery was observed.
  Duration of infusion was based on site clinical practice and the local package insert in both induction and consolidation periods.
  Maintenance period: Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once daily from days 1 to 28 in the maintenance period in C1 to 26 or a discontinuation criterion is met (1 cycle= 28 days).
  Interventions: Drug: Gilteritinib; Drug: Idarubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: Gilteritinib — Once-daily oral administration on 14 consecutive days in every cycle in each period.
  Other Names: Xospata; ASP2215
Drug: Idarubicin — Induction period: Once-daily intravenous injection of 12 mg/m^2 idarubicin on 3 consecutive days.
Drug: Cytarabine — Induction period: Once-daily intravenous injection of 100 mg/m^2 cytarabine on 7 consecutive days.
  Consolidation period: Twice-daily intravenous injection of 1.5 g/m^2 cytarabine on Days 1, 3, and 5.

SUMMARY:
The purpose of phase 1 part in this study was to determine the maximum tolerated dose (MTD) and/or recommended expansion dose (RED) of ASP2215 concomitant with cytarabine/idarubicin as induction chemotherapy based on the status of the onset of dose-limiting toxicity (DLT) in newly diagnosed Acute Myeloid Leukemia (AML) subjects. Phase 1 part also evaluated safety and tolerability and characterized the pharmacokinetic (PK) parameters of ASP2215 concomitant with induction and consolidation chemotherapy as well as evaluated the PK parameters of cytarabine concomitant with ASP2215.

The purpose of phase 2 part was to evaluate efficacy of ASP2215 in combination with induction therapy. Phase 2 cohort also evaluated safety and characterized the PK parameters of ASP2215 in combination with induction and consolidation therapy followed by maintenance therapy in newly diagnosed FLT3-mutated AML subjects.

DETAILED DESCRIPTION:
This study was composed of Phase 1 part (the dose-evaluation part and the expansion part) and Phase 2 part.

In the dose-evaluation part of Phase 1 part, at least 3 subjects received ASP2215 at each dose (low, middle, and high) for determination of MTD and/or RED. Treatment of AML in Phase 1 part was composed of 3 periods of therapy: remission induction, consolidation, and maintenance. The decision of whether or not to proceed to the next dose was made based on the occurrence of DLT during Cycle 1 of the induction period.

In the expansion part of Phase 1 part, a maximum of 3 subjects received ASP2215 at RED that had been recommended in the dose-evaluation part and the safety was assessed based on the onset of DLTs during Cycle 1 of the induction and consolidation periods.

In Phase 2 part, Subjects received ASP2215 at the recommended dose established in Phase 1 part. The target population was limited to newly diagnosed FLT3-mutated AML.

ELIGIBILITY:
Inclusion Criteria:

[Phase 1 part]

* Subject is defined as having previously untreated de novo AML according to the World Health Organization (WHO) criteria (2008) within 28 days prior to study enrollment.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Subject must meet all of the following criteria in the laboratory test at screening:

  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels of ≤ 2.5 × institutional upper limit of normal (ULN)
  * Total serum bilirubin level of ≤ 1.5 × institutional ULN
  * Serum creatinine level of ≤ 1.5 × institutional ULN or an estimated glomerular filtration rate (eGFR) of > 50 mL/min
* Subject is suitable for oral administration of ASP2215.
* Female subject falls under the following:

  * Of non-childbearing potential:
  * ・Post-menopausal (defined as at least 1 year with no menses without a medical reason such as drug administration) at screening, or
  * ・Documented surgically sterile or status post-hysterectomy (at least 1 month prior to screening)
  * Of childbearing potential:
  * ・Has a negative result for the pregnancy test at screening, and
  * ・Agrees to use an appropriate contraception starting at screening and throughout the study period and for 60 days after the final study drug administration
* Female subject agrees not to breastfeed starting at screening and throughout the study period and for 60 days after the final study drug administration.
* Female subject agrees not to donate ova starting at screening and throughout the study period and for 60 days after the final study drug administration.
* Male subject and his female spouse/partner who is of childbearing potential agrees to use an appropriate contraception starting at screening and throughout the study period and for 120 days after the final study drug administration.
* Male subject agrees not to donate sperm starting at screening and throughout the study period and for 120 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while on study treatment.
* Subject can be admitted during the induction period.

[Phase 2 part]

* Subject has a diagnosis of previously-untreated de novo acute myeloid leukemia (AML) according to World Health Organization (WHO) classification (2017) documented within 28 days prior to enrollment.
* Subject is positive for FLT3-ITD and/or TKD mutation in bone marrow or whole blood as determined by the central lab. Registration by the local lab result is not acceptable.
* Subject has an ECOG performance status (PS) 0 to 1. Subject who has an ECOG PS 2 is eligible only if the primary disease related symptoms such as pneumonia and febrile neutropenia are the cause of PS score.
* Subject is suitable for oral administration of ASP2215.
* Female subject is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 180 days after final study treatment administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 60 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 180 days after the final study drug administration.
* Male subject and their female partners who are of childbearing potential must be using highly effective contraception per locally accepted standards in addition to a barrier method starting at screening and continue throughout the study period and for 120 days after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for 120 days after the final study drug administration.
* Male subject with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 120 days after the final study treatment administration.
* Subject agrees not to participate in another interventional study while on treatment.
* Subject must meet the following criteria as indicated on the clinical laboratory tests:

  * Serum creatinine ≤ 1.5 × institutional upper limit of normal (ULN), or if serum creatinine outside normal range, then glomerular filtration rate (GFR) > 50 mL/min/1.73m^2 as calculated with the 4-parameter Modification of Diet in Renal Disease (MDRD) equation.
  * Serum total bilirubin ≤ 2.5 mg/dL (43 μmol/L), except for subjects with Gilbert's syndrome.
  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN. If liver abnormality by the primary disease is suspected, subject may be pre-registered to initiate the chemotherapy. Prior to registration, AST/ALT values must meet the criteria to continue the study.
  * Serum magnesium ≥ institutional lower limit of normal (LLN). Subject may pre-register without magnesium value, but subject must meet the criteria prior to the full registration on Day 8.
  * Serum potassium ≥ institutional lower limit of normal (LLN).

Exclusion Criteria:

[Phase 1 part]

* Subject was diagnosed with acute promyelocytic leukemia (APL).
* Subject has breakpoint cluster region-abelson (BCR-ABL)-positive leukemia (chronic myelogenous leukemia in blast crisis).
* Subject has active malignant tumors other than AML or myelodysplastic syndrome (MDS).
* Subject has received prior AML treatment except for the following:

  * Urgent leukapheresis
  * Hydroxyurea administration for emergency treatment of hyperleukocytosis (≤ 7 days)
  * Administration of retinoic acid before the diagnosis to exclude APL (≤ 7 days)
  * Supportive care using growth factors or cytokines
  * Steroid administration to treat hypersensitivity or blood transfusion reactions
* Subject has clinically active central nervous system leukemia.
* Subject has disseminated intravascular coagulation (DIC).
* Subject has had major surgery within 28 days prior to the first study drug administration.
* Subject has had radiation therapy within 28 days prior to the first study drug administration.
* Subject has congestive heart failure of New York Heart Association (NYHA) class 3 or 4, or subject with a past history of congestive heart failure of NYHA class 3 or 4 and in whom echocardiogram (ECHO) or Multiple Gate Acquisition (MUGA) scan performed within 3 months prior to screening or at screening showed a left ventricular ejection fraction (LVEF) of < 45%.
* Subject has cardiac impairment or a clinically significant cardiac disease, including any one of the following:

  * Complete left bundle branch block
  * Obligate use of a cardiac pacemaker
  * Long QT syndrome at Screening
  * Prolongation of the QTc interval (> 450 ms) on electrocardiogram (ECG) at screening
  * Right bundle branch block + left anterior hemiblock (bifascicular block)
  * Angina pectoris within 3 months prior to study drug administration
  * Acute myocardial infarction within 3 months prior to study drug administration
* Subject requires treatment with concomitant drugs that are strong inducers of cytochrome P450 (CYP)3A.
* Subject requires treatment with concomitant drugs that are strong inhibitors or inducers of P glycoprotein (P-gp) with the exception of drugs that are considered absolutely essential for the care of the subject.
* Subject requires treatment with concomitant drugs that target serotonin 5HT1 or 5HT2B receptors or sigma receptors, with the exception of drugs that are considered absolutely essential for treatment of the subject.
* Subject has an active uncontrollable infection.
* Subject is known to have human immunodeficiency virus (HIV) infection.
* Subject has active hepatitis B or C or other active hepatic disorders.
* Subject has any condition that, in the investigator's or sub-investigator's opinion, makes the subject unsuitable for study participation.
* Potassium and magnesium levels of below institutional lower limit of normal in the laboratory test at screening.

[Phase 2 part]

* Subject was diagnosed with acute promyelocytic leukemia (APL).
* Subject has known BCR-ABL-positive leukemia (chronic myelogenous leukemia in blast crisis).
* Subject has therapy-related AML.
* Subject has active malignant tumors other than AML.
* Subject has received previous therapy for AML, with the exception of the following:

  * Emergency leukapheresis
  * Emergency treatment for hyperleukocytosis with hydroxyurea for ≤ 10 days
  * Preemptive treatment with retinoic acid prior to exclusion of APL ≤ 7 days
  * Growth factor or cytokine support
  * Steroids for the treatment of hypersensitivity or transfusion reactions.
* Subject has QTcF interval > 450 ms (average of triplicate determinations based on central reading).
* Subject with long QT syndrome.
* Subject has clinically active central nervous system leukemia.
* Subject has had major surgery within 4 weeks prior to the first study dose.
* Subject has radiation therapy within 4 weeks prior to the first study dose.
* Subject has immediate life-threatening, severe complications of leukemia such as severe uncontrolled bleeding and/or severe disseminated intravascular coagulation
* Subject is known to have human immunodeficiency virus infection.
* Subject has active hepatitis B or C.
* Subject has an uncontrolled infection. An infection controlled with an approved or closely monitored antibiotic/antiviral/antifungal treatment is allowed.
* Subject has uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia, congestive heart failure New York Heart Association (NYHA) class 3 or 4 or subject has a history of congestive heart failure of NYHA class 3 or 4 and echocardiogram (ECHO) or Multiple Gate Acquisition (MUGA) scan performed within 3 months prior to screening or at screening showed a left ventricular ejection fraction (LVEF) of < 45%.
* Subject requires treatment with concomitant drugs that are strong inducers of cytochrome P450 (CYP) 3A.
* Subject requires treatment with concomitant drugs that target serotonin 5HT2B receptors or sigma nonspecific receptors, with the exception of drugs that are considered absolutely essential for treatment of the subject.
* Subject requires treatment with concomitant drugs that are strong inhibitors or inducers of P glycoprotein (P-gp) with the exception of drugs that are considered absolutely essential for the care of the subject.
* Subject has prior malignancies, except resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously will not be allowed.
* Subject has any condition which makes the subject unsuitable for study participation.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-02-26 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (55):
- Japan (45):
  - Site JP81037, Anjo, Aichi-ken
  - Site JP00003, Nagoya, Aichi-ken
  - Site JP81003, Nagoya, Aichi-ken
  - Site JP81027, Nagoya, Aichi-ken
  - Site JP81038, Toyohashi, Aichi-ken
  - Site JP81010, Narita, Chiba
  - Site JP81039, Matsuyama, Ehime
  - Site JP81007, Yoshida-gun, Fukui
  - Site JP00002, Maebashi, Gunma
  - Site JP81001, Maebashi, Gunma
  - Site JP81026, Fukuyama, Hiroshima
  - Site JP81018, Ōtake, Hiroshima
  - Site JP81014, Sapporo, Hokkaido
  - Site JP81015, Sapporo, Hokkaido
  - Site JP81043, Himeji, Hyōgo
  - Site JP00007, Kobe, Hyōgo
  - Site JP81006, Kobe, Hyōgo
  - Site JP81036, Mito, Ibaraki
  - Site JP81023, Tsukuba, Ibaraki
  - Site JP81020, Kanazawa, Ishikawa-ken
  - Site JP81013, Isehara, Kanagawa
  - Site JP00006, Yokohama, Kanagawa
  - Site JP81005, Yokohama, Kanagawa
  - Site JP81024, Yokohama, Kanagawa
  - Site JP81035, Sendai, Miyagi
  - SIte JP81011, Ōmura, Nagasaki
  - Site JP81041, Tenri, Nara
  - Site JP81022, Shimono, Tochigi
  - Site JP81040, Bunkyo-ku, Tokyo
  - Site JP00005, Shinagawa-ku, Tokyo
  - Site JP81032, Shinagawa-ku, Tokyo
  - Site JP81029, Akita
  - Site JP81008, Chiba
  - Site JP00001, Fukuoka
  - Site JP81004, Fukuoka
  - Site JP81025, Fukuoka
  - Site JP81031, Fukushima
  - Site JP81030, Gifu
  - Site JP81033, Kochi
  - Site JP81028, Kumamoto
  - Site JP81016, Kyoto
  - Site JP81012, Nagasaki
  - Site JP81009, Okayama
  - Site JP81019, Osaka
  - Site JP81021, Osaka
- South Korea (6):
  - Site KR82005, Busan
  - Site KR82002, Incheon
  - Site KR82001, Seoul
  - Site KR82003, Seoul
  - Site KR82004, Seoul
  - Site KR82006, Seoul
- Taiwan (4):
  - Site TW88604, Kaohsiung City
  - Site TW88602, Taichung
  - Site TW88601, Tainan
  - Site TW88603, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with newly diagnosed acute myeloid leukemia (AML) and participants newly diagnosed FMS-like tyrosine kinase-3, FMS-related tyrosine kinase 3 (FLT3)-mutated AML; were enrolled in Phase 1 and Phase 2, respectively.
Pre-assignment Details: Participants who met all inclusion criteria and none of the exclusion criteria were enrolled in the study.
Groups:
- Phase 1: Dose Evaluation (DEv): Induction period (IP):
  Participants received 120 milligrams (mg) gilteritinib (3 tablets of 40 mg) orally, once a day from days 4 to 17 in combination with chemotherapy (idarubicin: 12 milligrams per square meters per day [mg/m^2/day] on days 1 to 3, cytarabine: 100 mg/m^2/day on days 1 to 7) via intravenous (IV) infusion; in the induction period in cycles (C) 1 and 2 (1 cycle= 42 days). Duration of infusion was determined based on site clinical practice and the local package insert.
  Consolidation period (CP):
  Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 1 to 14 in combination with chemotherapy (cytarabine: 1500 mg/m^2, twice daily on days 1, 3, and 5) via IV infusion; in the consolidation period in C1 to 3 (1 cycle= 28 days). Duration of infusion was determined based on site clinical practice and the local package insert.
  Maintenance period (MP):
  Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 1 to 28 in the maintenance period in C1 to 26 or a discontinuation criterion is met (1 cycle= 28 days).
- Phase 1: Dose Expansion (DEx): Induction period:
  Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 4 to 17 in combination with chemotherapy (idarubicin: 12 mg/m^2/day on days 1 to 3, cytarabine: 100 mg/m^2/day on days 1 to 7) via IV infusion; in the induction period in C1 and 2 (1 cycle= 42 days). Duration of infusion was determined based on site clinical practice and the local package insert.
  Consolidation period:
  Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 1 to 14 in combination with chemotherapy (cytarabine: 1500 mg/m^2, twice daily on days 1, 3, and 5) via IV infusion; in the consolidation period in C1 to 3 (1 cycle= 28 days). Duration of infusion was determined based on site clinical practice and the local package insert.
  Maintenance period:
  Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 1 to 28 in the maintenance period in C1 to 26 or a discontinuation criterion is met (1 cycle= 28 days).
- Phase 2: FLT3-mutated AML: Induction period:
  Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 8 until blood recovery in combination with chemotherapy (idarubicin: 12 mg/m^2/day on days 1 to 3, cytarabine: 100 mg/m^2/day on days 1 to 7) via IV infusion; in the induction period in C1 and 2. Each cycle was allowed to be extended until blood recovery was observed. Duration of infusion was determined based on site clinical practice and the local package insert.
  Consolidation period:
  Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 1 until blood recovery in combination with chemotherapy (cytarabine: 1500 mg/m^2, twice daily on days 1, 3, and 5) via IV infusion; in the consolidation period in C1 to 3. Each cycle was allowed to be extended until blood recovery was observed. Duration of infusion was determined based on site clinical practice and the local package insert.
  Maintenance period:
  Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 1 to 28 in the maintenance period in C1 to 26 or a discontinuation criterion is met (1 cycle= 28 days).
Period: Phase 1(DEv):IP (2 Cycles;42 Days/Cycle)
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx) | Phase 2: FLT3-mutated AML
Started | 3 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Miscellaneous | 1 | 0 | 0
Period: Phase 1(DEv):CP (3 Cycles;28 Days/Cycle)
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx) | Phase 2: FLT3-mutated AML
Started | 2 | 0 | 0
Completed | 1 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Miscellaneous | 1 | 0 | 0
Period: Phase 1(DEv):MP(26 Cycles;28 Days/Cycle)
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx) | Phase 2: FLT3-mutated AML
Started | 1 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Miscellaneous | 1 | 0 | 0
Period: Phase 1(DEx):IP (2 Cycles;42 Days/Cycle)
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx) | Phase 2: FLT3-mutated AML
Started | 0 | 10 | 0
Completed | 0 | 3 | 0
Not Completed | 0 | 7 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Miscellaneous | 0 | 4 | 0
Not completed — There is no CR, CRp, or CRi after 2 Cycles of Therapy | 0 | 1 | 0
Not completed — Disease Relapse | 0 | 1 | 0
Period: Phase 1(DEx):CP (3 Cycles;28 Days/Cycle)
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx) | Phase 2: FLT3-mutated AML
Started | 0 | 3 | 0
Completed | 0 | 3 | 0
Not Completed | 0 | 0 | 0
Period: Phase 1(DEx):MP(26 Cycles;28 Days/Cycle)
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx) | Phase 2: FLT3-mutated AML
Started | 0 | 3 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 3 | 0
Not completed — Micellaneous | 0 | 3 | 0
Period: Phase 2:IP(2 Cycles;up to 56 Days/Cycle)
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx) | Phase 2: FLT3-mutated AML
Started | 0 | 0 | 84
Completed | 0 | 0 | 62
Not Completed | 0 | 0 | 22
Not completed — Miscellaneous | 0 | 0 | 2
Not completed — Disease Relapse | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Lack of Efficacy | 0 | 0 | 3
Not completed — Death | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 2
Period: Phase 2:CP(4 Cycles;up to 28 Days/Cycle)
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx) | Phase 2: FLT3-mutated AML
Started | 0 | 0 | 57
Completed | 0 | 0 | 42
Not Completed | 0 | 0 | 15
Not completed — Miscellaneous | 0 | 0 | 7
Not completed — Disease Relapse | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 4
Period: Phase 2:MP(26 Cycles; 28 Days/Cycle)
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx) | Phase 2: FLT3-mutated AML
Started | 0 | 0 | 46
Completed | 0 | 0 | 23
Not Completed | 0 | 0 | 23
Not completed — Disease relapse | 0 | 0 | 11
Not completed — Miscellaneous | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Death | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF): All participants who received at least 1 dose of study drug were included.
Groups:
- Phase 1: Dose Evaluation (DEv); Phase 1: Dose Expansion (DEx): Induction period:
  Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 4 to 17 in combination with chemotherapy (idarubicin: 12 mg/m^2/day on days 1 to 3, cytarabine: 100 mg/m^2/day on days 1 to 7) via IV infusion; in the induction period in C1 and 2 (1 cycle= 42 days). Duration of infusion was determined based on site clinical practice and the local package insert.
  Consolidation period:
  Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 1 to 14 in combination with chemotherapy (cytarabine: 1500 mg/m^2, twice daily on days 1, 3, and 5) via IV infusion; in the consolidation period in C1 to 3 (1 cycle= 28 days). Duration of infusion was determined based on site clinical practice and the local package insert.
  Maintenance period:
  Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 1 to 28 in the maintenance period in C1 to 26 or a discontinuation criterion is met (1 cycle= 28 days).
- Total: Total of all reporting groups
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx) | Phase 2: FLT3-mutated AML | Total
Number analyzed (Participants) | 3 | 10 | 84 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.3 (14) | 49.9 (15) | 51 (14.4) | 50.8 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 43 | 48
  Male | 1 | 7 | 41 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 10 | 84 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 10 | 84 | 97
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 Part: Maximum Tolerated Dose (MTD) of Gilteritinib
Description: The MTD was defined as the highest dose of gilteritinib at which the posterior mean of the DLT incidence during Cycle 1 of induction therapy was estimated to be closest to 33%.
Time Frame: Day 1 up to the end of Induction period cycle 1 (up to 42 days)
Population: Dose-Determining Analysis Set (DDAS) Phase 1 part: Participants who received more than 80% of the intended dose of gilteritinib and safety was adequately assessed during DLT assessment period specified in each part were included.
Measure: Number; unit: miligram (mg)
Arm/Group | Phase 1: Dose Evaluation (DEv)
Number analyzed (Participants) | 3
miligram (mg) | NA — The posterior mean of DLT incidence estimated was lower than the pre-specified value of 33%, therefore, MTD was not reached.

2. Primary Outcome: Phase 1 Part: Recommended Expansion Dose (RED) of Gilteritinib
Description: RED was the recommended dose used in Phase 2 of the study that was decided by the sponsor's responsible person by comprehensively assessing the data obtained from the study.
Time Frame: Day 1 up to the end of Induction period cycle 1 (up to 42 days)
Population: Participants in the DDAS.
Measure: Number; unit: mg
Arm/Group | Phase 1: Dose Evaluation (DEv)
Number analyzed (Participants) | 3
mg | 120

3. Primary Outcome: Phase 1 Part: Number of Participants With Dose Limiting Toxicities (DLTs) of Gilteritinib
Description: DLTs were defined as:
  Any Grade ≥ 3 non-hematologic or extramedullary toxicity with the following exceptions:
  * Anorexia or fatigue
  * Grade 3 nausea and/or vomiting if participant did not require tube feeding or total parenteral nutrition, or diarrhea if the events did not require or prolong hospitalization that could be managed to grade ≤ 2 with standard antiemetic or antidiarrheal medications used at prescribed dose within 7 days of onset.
  * Grade 3 mucositis that resolved to Grade ≤ 2 within 7 days of onset, fever with neutropenia, with or without infection, infection
  * Grade 4 peripheral neutrophil count < 500/cubic millimeters (mm^3)
  * Platelet count < 20,000/mm^3 due to bone marrow hypoplasia
  * Grade ≥ 3 platelet count < 50,000/mm^3 accompanying bleeding
  * Grade 4 platelet count < 25,000/mm^3 requiring platelet transfusion
  DLT was assessed until cycle 1 of dose evaluation induction period and until cycle 1 of dose expansion consolidation period.
Time Frame: Day 1 up to the end of Consolidation Cycle 1 (approximately up to 4 months)
Population: Participants in the DDAS.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx)
Number analyzed (Participants) | 3 | 10
Participants | 0 | 1

4. Primary Outcome: Phase 1 Part: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE could therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. TEAE included both serious and non-serious AEs. TEAE for Phase 1 was defined as an AE observed after the date of first dose until 30 days after the last dose.
Time Frame: From the date of first dose up to 30 days after the last dose ( maximum duration up to approximately 4.1 years)
Population: SAF
Measure: Number; unit: Participants
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx)
Number analyzed (Participants) | 3 | 10
Participants | 3 | 10

5. Primary Outcome: Phase 2 Part: Complete Remission (CR) Rate: Induction Period
Description: Percentage of participants with CR was reported. CR was defined as a morphologically leukemia-free state at the post-baseline visit, having a neutrophil count of ≥ 1,000/mm3 and platelet count of ≥ 100,000/mm3, bone marrow blasts < 5%. No evidence of Auer rods and no evidence of extramedullary leukemia. The blast counts in peripheral blood was ≤ 2%.
Time Frame: From the date of first dose up to the start of Consolidation (approximately up to 4 months)
Population: Participants in the Full Analysis Set (FAS) Phase 2 part: Participants who received at least 1 dose of study drug and had at least one post-baseline bone marrow assessment were included.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 82
Percentage of participants | 50 [40.4 to 59.6]

6. Secondary Outcome: Phase 1 Part: Maximum Concentration (Cmax) of Gilteritinib Concomitant With Induction and Consolidation Chemotherapy
Description: Cmax was derived from the PK samples collected. It was planned that standard deviation(SD) would only be calculated if there are more than 3 participants analyzed otherwise, SD was not calculated.
Time Frame: Induction period: Pre-dose, 1, 2, 4, 6, 10, and 24 hours post-dose on Cycle 1 Day 4 Consolidation period: Pre-dose, 1, 2, 4, 6, 10, and 24 hours post-dose on Cycle 1 Day 1
Population: Pharmacokinetics Analysis Set (PKAS): Participants who received the study drug, from whom samples for drug concentration measurement were collected for at least 1 time-point after the study drug administration, and from whom drug concentration measurement was obtained were included. PKAS with available data analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx)
Number analyzed (Participants) | 3 | 10
nanograms per milliliter (ng/mL)
  Induction Period | 246 (154) | 132 (27.5)
  Consolidation period: number analyzed (Participants) | 2 | 3
  Consolidation period | 133 (NA) — Since there were less than 3 participants analyzed, SD was not calculated nor reported. | 73.5 (17.5)

7. Secondary Outcome: Phase 1 Part: Time to Attain Cmax (Tmax) of Gilteritinib Concomitant With Induction and Consolidation Chemotherapy
Description: Tmax was derived from the PK samples collected.
Time Frame: as for outcome 6
Population: PKAS with available data analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx)
Number analyzed (Participants) | 3 | 10
hours
  Induction period | 3.93 [3.82 to 6.13] | 5.77 [3.83 to 9.77]
  Consolidation period: number analyzed (Participants) | 2 | 3
  Consolidation period | 2.94 [1.85 to 4.03] | 4.32 [3.90 to 9.70]

8. Secondary Outcome: Phase 1 Part: Area Under Plasma Concentration-time Curve From Time 0 to 24 (AUC24) of Gilteritinib Concomitant With Induction and Consolidation Chemotherapy
Description: AUC24 was derived from the PK samples collected. It was planned that standard deviation(SD) would only be calculated if there are more than 3 participants analyzed otherwise, SD was not calculated.
Time Frame: as for outcome 6
Population: PKAS with available data analyzed.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx)
Number analyzed (Participants) | 3 | 10
ng*hr/mL
  Induction period | 3880 (2530) | 2210 (567)
  Consolidation period: number analyzed (Participants) | 2 | 3
  Consolidation period | 2110 (NA) — Since there were less than 3 participants analyzed, SD was not calculated nor reported. | 1160 (204)

9. Secondary Outcome: Phase 1 Part: Area Under The Concentration-Time Curve From The Time Zero to The Last Measurable Concentration (AUClast) of Gilteritinib Concomitant With Induction and Consolidation Chemotherapy
Description: AUClast was derived from the PK samples collected. It was planned that standard deviation(SD) would only be calculated if there are more than 3 participants analyzed otherwise, SD was not calculated.
Time Frame: as for outcome 6
Population: PKAS with available data analyzed.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Phase 1: Dose Expansion (DEx): Induction period:
  Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day from days 4 to 17 in combination with chemotherapy (idarubicin: 12 mg/m^2/day on days 1 to 3, cytarabine: 100 mg/m^2/day on days 1 to 7) via IV infusion; in the induction period in C1 and 2 (1 cycle= 42 days). Duration of infusion was determined based on site clinical practice and the local package insert.
  Consolidation period:
  Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day from days 1 to 14 in combination with chemotherapy (cytarabine: 1500 mg/m^2, twice daily on days 1, 3, and 5) via IV infusion; in the consolidation period in C1 to 3 (1 cycle= 28 days). Duration of infusion was determined based on site clinical practice and the local package insert.
  Maintenance period:
  Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day from days 1 to 28 in the maintenance period in C1 to 26 or a discontinuation criterion is met (1 cycle= 28 days).
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx)
Number analyzed (Participants) | 3 | 10
ng*hr/mL
  Induction period | 3830 (2520) | 2190 (552)
  Consolidation period: number analyzed (Participants) | 2 | 3
  Consolidation period | 2090 (NA) — Since there were less than 3 participants analyzed, SD was not calculated nor reported. | 1150 (202)

10. Secondary Outcome: Phase 1 Part: Plasma Trough Concentration (Ctrough) of Gilteritinib Concomitant With Induction and Consolidation Chemotherapy
Description: Ctrough is the plasma concentration prior to drug administration. It was planned that standard deviation(SD) would only be calculated if there are more than 3 participants analyzed otherwise, SD was not calculated.
Time Frame: Induction period: Pre-dose on Cycle 1 Day 8, 11, and 17 Consolidation period: Pre-dose on Cycle 1 Day 6 and 15
Population: PKAS with available data analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx)
Number analyzed (Participants) | 3 | 9
ng/mL
  Induction period: Cycle 1 day 8 | 245 (144) | 245 (77.7)
  Induction period: Cycle 1 day 11 | 283 (183) | 417 (203)
  Induction period: Cycle 1 day 17: number analyzed (Participants) | 3 | 8
  Induction period: Cycle 1 day 17 | 393 (252) | 455 (143)
  Consolidation period: Cycle 1 day 6: number analyzed (Participants) | 2 | 3
  Consolidation period: Cycle 1 day 6 | 194 (NA) — Since there were less than 3 participants analyzed, SD was not calculated nor reported. | 159 (12.1)
  Consolidation period: Cycle 1 day 15: number analyzed (Participants) | 2 | 3
  Consolidation period: Cycle 1 day 15 | 285 (NA) — Since there were less than 3 participants analyzed, SD was not calculated nor reported. | 171 (154)

11. Secondary Outcome: Phase 1 Part: Plasma Trough Concentration of Cytarabine Concomitant With Gilteritinib With Induction and Consolidation Period
Description: as for outcome 10
Time Frame: Induction period: Predose on Cycle 1 Day 1, 3, and 8 Consolidation period: Predose on Cycle 1 Day 2 and 6
Population: PKAS with available data analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx)
Number analyzed (Participants) | 3 | 9
ng/mL
  Induction period: Cycle 1 Day 1: number analyzed (Participants) | 3 | 7
  Induction period: Cycle 1 Day 1 | 0 (NA) — Since the mean concentration of pre-dose of Cytarabine is zero, therefore, SD was not estimated. | 0 (NA) — Since the mean concentration of pre-dose of Cytarabine is zero, therefore, SD was not estimated.
  Induction period: Cycle 1 Day 3: number analyzed (Participants) | 3 | 6
  Induction period: Cycle 1 Day 3 | 34.9 (14.5) | 210 (417)
  Induction period: Cycle 1 Day 8 | 58.8 (8.67) | 110 (107)
  Consolidation period: Cycle 1 Day 2: number analyzed (Participants) | 2 | 3
  Consolidation period: Cycle 1 Day 2 | 4.87 (NA) — Since there were less than 3 participants analyzed, SD was not calculated nor reported. | 9.39 (2.19)
  Consolidation period: Cycle 1 Day 6: number analyzed (Participants) | 2 | 3
  Consolidation period: Cycle 1 Day 6 | 7.09 (NA) — Since there were less than 3 participants analyzed, SD was not calculated nor reported. | 11.8 (1.91)

12. Secondary Outcome: Phase 2 Part: Plasma Trough Concentration of Gilteritinib Concomitant With Induction and Consolidation Chemotherapy
Description: Ctrough is the plasma concentration prior to drug administration.
Time Frame: Induction period : Predose on Cycle 1 Day 15 and 21 Consolidation period: Predose on Cycle 1 Day 8 and 15
Population: PKAS with available data analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 83
ng/mL
  Induction Period: Cycle 1 Day 15 | 522 (331)
  Induction Period: Cycle 1 Day 21: number analyzed (Participants) | 80
  Induction Period: Cycle 1 Day 21 | 647 (518)
  Consolidation Period: Cycle 1 Day 8: number analyzed (Participants) | 55
  Consolidation Period: Cycle 1 Day 8 | 244 (152)
  Consolidation Period: Cycle 1 Day 15: number analyzed (Participants) | 57
  Consolidation Period: Cycle 1 Day 15 | 375 (249)

13. Secondary Outcome: Phase 2 Part: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from the date of first dose of day 1 to the date of death due to any cause. Participants still alive or lost to follow up was censored at the time they were last known to be alive. Kaplan-Meier (KM) estimate was used for analysis.
Time Frame: From the date of first dose up to the date of death (maximum duration: approximately 4.4 years)
Population: Time-to-Event-FAS (TTE-FAS): All participants who received at least 1 dose of gilteritinib with or without postbaseline bone marrow assessments.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 84
Months | 48.2 [45.1 to NA] — The upper limit of the confidence interval of the median survival time was not estimable, since the upper limit of the confidence interval of the Kaplan-Meier plot did not reach 50% survival due to insufficient number of events.

14. Secondary Outcome: Phase 2 Part: Event Free Survival (EFS)
Description: Event-free survival (EFS): time from date of first dose of study regimen until date of documented relapse, treatment failure or death from any cause, whichever occurred first. KM estimate was used for analysis. Relapse: reappearance of leukemic blasts in peripheral blood (>2%)/≥ 5% blasts in bone marrow aspirate (BMA)/reappearance of significant numbers of peripheral blasts and an increase in percentage of blasts in BMA to > 25%. Treatment failure: participants who failed to achieve composite complete remission (CRc) or who discontinued treatment due to "lack of efficacy" without previous response. CRc: rate of all complete & incomplete remissions i.e. CR + CR with incomplete platelet recovery (CRp) + CR with incomplete hematological recover (CRi). CRp: met all CR criteria at post-baseline visit, except unrecovered platelet count (< 100,000/mm^3). CRi: met all CR criteria at post-baseline visit, except unrecovered neutrophil count (< 1,000/mm^3). CR: defined in outcome measure #5.
Time Frame: From the date of first dose up to the date of documented relapse, treatment failure or death from any cause (maximum duration: approximately 4.4 years)
Population: TTE-FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 84
Months | 25.0 [11.3 to 48.2]

15. Secondary Outcome: Phase 2 Part: Relapse Free Survival (RFS)
Description: Relapse-free survival (RFS): time from date of achievement of first CRc until relapse or death from any cause. KM estimate was used for analysis.
  Relapse: reappearance of leukemic blasts in peripheral blood (>2%)/≥ 5% blasts in bone marrow aspirate (BMA)/reappearance of significant numbers of peripheral blasts and an increase in percentage of blasts in BMA to > 25%.
  CRc: rate of all complete & incomplete remissions i.e. CR + CR with incomplete platelet recovery (CRp) + CR with incomplete hematological recover (CRi).
  CRp: met all CR criteria at post-baseline visit, except unrecovered platelet count (< 100,000/mm^3).
  CRi: met all CR criteria at post-baseline visit, except unrecovered neutrophil count (< 1,000/mm^3).
  CR: morphologically leukemia-free state at post-baseline visit, having neutrophil count of ≥ 1,000/mm^3 and platelet count of ≥ 100,000/mm^3, bone marrow blasts < 5%. No evidence of Auer rods & extramedullary leukemia. Blast counts in peripheral blood was ≤ 2%.
Time Frame: From the date of achievement of first CRc up to the date of documented relapse or death from any cause (maximum duration: approximately 3.9 years)
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 82
Months | 27.8 [17.4 to 39.8]

16. Secondary Outcome: Phase 2 Part: CR Rate After Consolidation and Maintenance Period
Description: Percentage of participants with CR was reported. CR was defined as a morphologically leukemia-free state at the post-baseline visit, having a neutrophil count of ≥ 1,000/mm^3 and platelet count of ≥ 100,000/mm^3, bone marrow blasts < 5%. No evidence of Auer rods and no evidence of extramedullary leukemia. The blast counts in peripheral blood was ≤ 2%. Derived response assessment after the consolidation period refers to the best response from the start of treatment in the induction period until the end of the consolidation period and for the maintenance period refers to the best response from the start of treatment in the induction period until the end of the maintenance period.
Time Frame: CP: From date of first dose up to end of period (approximately 1.8 years), MP: From date of first dose up to the end of period (approximately 3.8 years)
Population: The analysis population consisted of FAS participants, regardless of whether they proceeded to consolidation or maintenance. CR rate after consolidation included participants from induction through consolidation and CR rate after maintenance included participants from induction through maintenance.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 82
Percentage of participants
  After consolidation period | 63.4 [52.0 to 73.8]
  After maintenance period | 63.4 [52.0 to 73.8]

17. Secondary Outcome: Phase 2 Part: CR Rate Without Minimal Residual Disease (MRD) After Each Treatment Therapy Period
Description: CR% without MRD reported. CR rate without MRD after each treatment therapy was defined similarly as CR rate after each treatment therapy. Responders achieve that the best response is CR and MRD status was negative. CR was defined as a morphologically leukemia-free state, having a neutrophil count of ≥ 1,000/mm^3 and platelet count of ≥ 100,000/mm^3, bone marrow blasts < 5%. No evidence of Auer rods and extramedullary leukemia. The blast counts in peripheral blood was ≤ 2%. Derived response assessment after the IP refers to the best response from the start of treatment in the IP until the end of the IP, after CP refers to the best response from the start of treatment in the IP until the end of the CP and for the MP refers to the best response from the start of treatment in the IP until the end of the MP.
Time Frame: IP: From date of first dose up to end of period (approximately 1.4 years), CP: From date of first dose up to end of period (approximately 1.8 years), MP: From date of first dose up to the end of period (approximately 3.8 years)
Population: The analysis population consisted of FAS participants, regardless of whether they proceeded to induction, consolidation or maintenance. CR rate after: induction included participants from start of treatment through induction; consolidation included participants from induction through consolidation and maintenance included participants from induction through maintenance.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 82
Percentage of participants
  After Induction Period | 18.3 [10.6 to 28.4]
  After Consolidation Period | 35.4 [25.1 to 46.7]
  After Maintenance Period | 35.4 [25.1 to 46.7]

18. Secondary Outcome: Phase 2 Part: CR With Partial Hematological Recovery (CRh) Rate After Each Treatment Therapy Period
Description: Percentage of participants with CRh was reported. CRh was defined as a condition at the post baseline visit, having bone marrow blasts < 5%, partial hematologic recovery neutrophil count≥ 500/mm^3 and platelet count ≥ 50,000/mm^3, no evidence of extramedullary leukemia and could be classified as CR. The blast counts in peripheral blood was ≤ 2%. Derived response assessment after the IP refers to the best response from the start of treatment in the IP until the end of the IP, after CP refers to the best response from the start of treatment in the IP until the end of the CP and for the MP refers to the best response from the start of treatment in the IP until the end of the MP.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Phase 2: FLT3-mutated AML: Induction period:
  Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 8 until blood recovery in combination with chemotherapy (idarubicin: 12 mg/m^2/day on days 1 to 3, cytarabine: 100 mg/m^2/day on days 1 to 7) via IV infusion; in the induction period in C1 and 2. Each cycle was allowed to be extended until blood recovery was observed. Duration of infusion was determined based on site clinical practice and the local package insert.
  Consolidation period:
  Participants received 120 mg gilteritinib (3 tablets of 40 mg) orally, once a day from days 1 until blood recovery in combination with chemotherapy (cytarabine: 1500 mg/m^2, twice daily on days 1, 3, and 5) via IV infusion; in the consolidation period in C1 to 3. Each cycle was allowed to be extended until blood recovery was observed. Duration of infusion was determined based on site clinical practice and the local package insert.
  Maintenance period:
  Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day from days 1 to 28 in the maintenance period in C1 to 26 or a discontinuation criterion is met (1 cycle= 28 days).
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 82
Percentage of participants
  After Induction Period | 17.1 [9.7 to 27.0]
  After Consolidation Period | 9.8 [4.3 to 18.3]
  After Maintenance Period | 9.8 [4.3 to 18.3]

19. Secondary Outcome: Phase 2 Part: Composite CR (CRc) Rate After Each Treatment Therapy Period
Description: Percentage of participants with CRc reported. CRc: rate of all complete & incomplete remissions i.e. CR + CR with incomplete platelet recovery (CRp) + CR with incomplete hematological recovery (CRi). CRp: met all CR criteria, except unrecovered platelet count (< 100,000/mm^3). CRi: met all CR criteria, except unrecovered neutrophil count (< 1,000/mm^3). CR: morphologically leukemia-free state, having neutrophil count of ≥ 1,000/mm^3 and platelet count of ≥ 100,000/mm^3, bone marrow blasts < 5%. No evidence of Auer rods & extramedullary leukemia. Blast counts in peripheral blood was ≤ 2%. Derived response assessment after the IP refers to the best response from the start of treatment in the IP until the end of the IP, after CP refers to the best response from the start of treatment in the IP until the end of the CP and for the MP refers to the best response from the start of treatment in the IP until the end of the MP.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 82
Percentage of participants
  After Induction Period | 86.6 [77.3 to 93.1]
  After Consolidation Period | 87.8 [78.7 to 94.0]
  After Maintenance Period | 87.8 [78.7 to 94.0]

20. Secondary Outcome: Phase 2 Part: CR/CRh Rate After Each Treatment Therapy Period
Description: Percentage of participants with CR/CRh was reported. CR was defined as a morphologically leukemia-free state at the post-baseline visit, having a neutrophil count of ≥ 1,000/mm^3 and platelet count of ≥ 100,000/mm^3, bone marrow blasts < 5%. No evidence of Auer rods and no evidence of extramedullary leukemia. The blast counts in peripheral blood was ≤ 2%. CRh was defined as a condition at the post baseline visit, having bone marrow blasts < 5%, partial hematologic recovery neutrophil count≥ 500/mm^3 and platelet count ≥ 50,000/mm^3, no evidence of extramedullary leukemia and could be classified as CR. The blast counts in peripheral blood was ≤ 2%. Derived response assessment after the IP refers to the best response from the start of treatment in the IP until the end of the IP, after CP refers to the best response from the start of treatment in the IP until the end of the CP and for the MP refers to the best response from the start of treatment in the IP until the end of the MP.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 82
Percentage of participants
  After Induction Period | 67.1 [55.8 to 77.1]
  After Consolidation Period | 73.2 [62.2 to 82.4]
  After Maintenance Period | 73.2 [62.2 to 82.4]

21. Secondary Outcome: Phase 2 Part: Duration of CR
Description: Duration of CR was defined as the time from the date of achieving first CR until the date of first documented relapse for participants who achieved CR. KM estimate was used for analysis.
  CR was defined as a morphologically leukemia-free state at the post-baseline visit, having a neutrophil count of ≥ 1,000/mm^3 and platelet count of ≥ 100,000/mm^3, bone marrow blasts < 5%. No evidence of Auer rods and no evidence of extramedullary leukemia. The blast counts in peripheral blood was ≤ 2%.
  Relapse: reappearance of leukemic blasts in peripheral blood (>2%)/≥ 5% blasts in BMA/reappearance of numbers of peripheral blasts and an increase in percentage of blasts in BMA to > 25%.
Time Frame: From the date of achieving CR up to the date of documented relapse (maximum duration: approximately 2.6 years)
Population: FAS with available data analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 55
Months | NA [NA to NA] — The median survival time and the upper/lower limits of the confidence interval of median survival time were not estimable, since the KM plot and its upper/lower limit of the confidence interval did not reach 50% survival due to insufficient number of events.

22. Secondary Outcome: Phase 2 Part: Duration of CR/CRh
Description: Duration of CR/CRh is defined as the time from the date of achieving first CR/CRh until the date of first documented relapse for participants who achieved CR/CRh. KM estimate was used for analysis. CR was defined as a morphologically leukemia-free state at the post-baseline visit, having a neutrophil count of ≥ 1,000/mm^3 and platelet count of ≥ 100,000/mm^3, bone marrow blasts < 5%. No evidence of Auer rods and no evidence of extramedullary leukemia. The blast counts in peripheral blood was ≤ 2%. CRh was defined as a condition at the post baseline visit, having bone marrow blasts < 5%, partial hematologic recovery neutrophil count≥ 500/mm^3 and platelet count ≥ 50,000/mm^3, no evidence of extramedullary leukemia and could be classified as CR. The blast counts in peripheral blood was ≤ 2%.
  Relapse: reappearance of leukemic blasts in peripheral blood (>2%)/≥ 5% blasts in BMA/reappearance of numbers of peripheral blasts and an increase in percentage of blasts in BMA to > 25%.
Time Frame: From the date of achieving CR/CRh up to the date of documented relapse (maximum duration: approximately 2.6 years)
Population: FAS with available data analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 63
Months | NA [NA to NA] — The median survival time and the upper/lower limits of the confidence interval of median survival time were not estimable, since the KM plot and its upper/lower limit of the confidence interval did not reach 50% survival due to insufficient number of events.

23. Secondary Outcome: Phase 2 Part: Duration of CRh
Description: Duration of CRh was defined as the time from date of achieving first CRh until date of first documented relapse for participants who achieved CRh. KM estimate was used for analysis. CRh was defined as a condition at the post baseline visit, having bone marrow blasts < 5%, partial hematologic recovery neutrophil count≥ 500/mm^3 and platelet count ≥ 50,000/mm^3, no evidence of extramedullary leukemia and could be classified as CR. The blast counts in peripheral blood was ≤ 2%.
  Relapse: reappearance of leukemic blasts in peripheral blood (>2%)/≥ 5% blasts in BMA/reappearance of numbers of peripheral blasts and an increase in percentage of blasts in BMA to > 25%.
Time Frame: From the date of achieving CRh up to the date of documented relapse (maximum duration: approximately 2.6 years)
Population: FAS with available data analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 45
Months | NA [NA to NA] — The median survival time and the upper/lower limits of the confidence interval of median survival time were not estimable, since the KM plot and its upper/lower limit of the confidence interval did not reach 50% survival due to insufficient number of events.

24. Secondary Outcome: Phase 2 Part: Duration of CRc
Description: Duration of CRc is defined as the time from the date of achieving first CRc until the date of first documented relapse for participants who achieved CRc. KM estimate was used for analysis. CRc: rate of all complete & incomplete remissions i.e. CR + CR with incomplete platelet recovery (CRp) + CR with incomplete hematological recover (CRi). CRp: met all CR criteria at post-baseline visit, except unrecovered platelet count (< 100,000/mm^3). CRi: met all CR criteria at post-baseline visit, except unrecovered neutrophil count (< 1,000/mm^3). CR: morphologically leukemia-free state at post-baseline visit, having neutrophil count of ≥ 1,000/mm^3 and platelet count of ≥ 100,000/mm^3, bone marrow blasts < 5%. No evidence of Auer rods & extramedullary leukemia. Blast counts in peripheral blood was ≤ 2%.
  Relapse: reappearance of leukemic blasts in peripheral blood (>2%)/≥ 5% blasts in BMA/reappearance of numbers of peripheral blasts and an increase in percentage of blasts in BMA to > 25%.
Time Frame: From the date of achieving CRc up to the date of documented relapse (maximum duration: approximately 2.7 years)
Population: FAS with available data analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 75
Months | NA [NA to NA] — The median survival time and the upper/lower limits of the confidence interval of median survival time were not estimable, since the KM plot and its upper/lower limit of the confidence interval did not reach 50% survival due to insufficient number of events.

25. Secondary Outcome: Phase 2 Part: Duration of Response (DoR)
Description: DoR: from first day of achieving CRc (CR+ CRp,+CRi)/partial remission (PR) to first day of relapse. KM estimate was used for analysis. CR: morphologically leukemia-free state at post-baseline visit, having neutrophil count of ≥ 1,000/mm^3 & platelet count of ≥ 100,000/mm^3, bone marrow blasts < 5%. No evidence of Auer rods & extramedullary leukemia. Peripheral blood blast counts was ≤ 2%. CRp: met all CR criteria at post-baseline visit, except unrecovered platelet count (< 100,000/mm^3). CRi: met all CR criteria at post-baseline visit, except unrecovered neutrophil count (< 1,000/mm^3). PR: condition with regeneration of normal hematopoietic cells in bone marrow, no detectable blasts, ≥ 50% decrease of blasts in BMA & total bone marrow blasts of 5-25%. No evidence of extramedullary leukemia. Relapse: reappearance of leukemic blasts in peripheral blood (>2%)/≥ 5% blasts in BMA/reappearance of numbers of peripheral blasts and an increase in percentage of blasts in BMA to > 25%
Time Frame: From the date of achieving CR, CRp, CRi/PR up to the date of documented relapse (maximum duration: approximately 2.7 years)
Population: FAS with available data analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 76
Months | NA [NA to NA] — The median survival time and the upper/lower limits of the confidence interval of median survival time were not estimable, since the KM plot and its upper/lower limit of the confidence interval did not reach 50% survival due to insufficient number of events.

26. Secondary Outcome: Phase 2 Part: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE could therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. TEAE for Phase 2 was defined as an AE observed after the date of first dose until 30 days after the last dose. TEAE included both serious and non-serious AEs.
Time Frame: From the date of first dose up to 30 days after the last dose ( maximum duration up to approximately 4.4 years)
Population: SAF
Measure: Number; unit: Participants
Arm/Group | Phase 2: FLT3-mutated AML
Number analyzed (Participants) | 84
Participants | 84

ADVERSE EVENTS:
Time Frame: Adverse events: Phase 1: From the date of first dose up to 30 days after the last dose ( maximum duration up to approximately 4.1 years) Phase 2: From the date of first dose up to 30 days after the last dose ( maximum duration up to approximately 4.4 years) All-cause mortality: From randomization up to approximately 9.4 years.
Description: SAF
Groups:
- Phase 1: Dose Evaluation (DEv): Induction period (IP):
  Participants received 120 milligrams (mg) giltertinib (3 tablets of 40 mg) orally, once a day from days 4 to 17 in combination with chemotherapy (idarubicin: 12 milligrams per square meters per day [mg/m^2/day] on days 1 to 3, cytarabine: 100 mg/m^2/day on days 1 to 7) via intravenous (IV) infusion; in the induction period in cycles (C) 1 and 2 (1 cycle= 42 days). Duration of infusion was determined based on site clinical practice and the local package insert.
  Consolidation period (CP):
  Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day from days 1 to 14 in combination with chemotherapy (cytarabine: 1500 mg/m^2, twice daily on days 1, 3, and 5) via IV infusion; in the consolidation period in C1 to 3 (1 cycle= 28 days). Duration of infusion was determined based on site clinical practice and the local package insert.
  Maintenance period (MP):
  Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day from days 1 to 28 in the maintenance period in C1 to 26 or a discontinuation criterion is met (1 cycle= 28 days).
- Phase 1: Dose Expansion (DEx): Induction period (IP):
  Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day from days 4 to 17 in combination with chemotherapy (idarubicin: 12 mg/m^2/day on days 1 to 3, cytarabine: 100 mg/m^2/day on days 1 to 7) via IV infusion; in the induction period in C1 and 2 (1 cycle= 42 days). Duration of infusion was determined based on site clinical practice and the local package insert.
  Consolidation period (CP):
  Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day from days 1 to 14 in combination with chemotherapy (cytarabine: 1500 mg/m^2, twice daily on days 1, 3, and 5) via IV infusion; in the consolidation period in C1 to 3 (1 cycle= 28 days). Duration of infusion was determined based on site clinical practice and the local package insert.
  Maintenance period (MP):
  Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day from days 1 to 28 in the maintenance period in C1 to 26 or a discontinuation criterion is met (1 cycle= 28 days).
- Phase 2: FLT3-mutated AML: Induction period (IP):
  Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day from days 8 until blood recovery in combination with chemotherapy (idarubicin: 12 mg/m^2/day on days 1 to 3, cytarabine: 100 mg/m^2/day on days 1 to 7) via IV infusion; in the induction period in C1 and 2. Each cycle was allowed to be extended until blood recovery was observed. Duration of infusion was determined based on site clinical practice and the local package insert.
  Consolidation period (CP):
  Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day from days 1 until blood recovery in combination with chemotherapy (cytarabine: 1500 mg/m^2, twice daily on days 1, 3, and 5) via IV infusion; in the consolidation period in C1 to 3. Each cycle was allowed to be extended until blood recovery was observed. Duration of infusion was determined based on site clinical practice and the local package insert.
  Maintenance period (MP):
  Participants received 120 mg giltertinib (3 tablets of 40 mg) orally, once a day from days 1 to 28 in the maintenance period in C1 to 26 or a discontinuation criterion is met (1 cycle= 28 days).
Arm/Group | Phase 1: Dose Evaluation (DEv) | Phase 1: Dose Expansion (DEx) | Phase 2: FLT3-mutated AML
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/10 | 25/84
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/10 | 45/84
Other Adverse Events (participants affected / at risk) | 3/3 | 10/10 | 84/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Evaluation (DEv) (N=3) | Phase 1: Dose Expansion (DEx) (N=10) | Phase 2: FLT3-mutated AML (N=84)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (7)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 3 (5)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 4 (4)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 6 (10)
Acute graft versus host disease (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Graft versus host disease (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 9 (12)
Root canal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 9 (11)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 3 (4)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Splenic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Liver function test abnormal (Investigations) | 1 (2) | 1 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (4)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acquired antithrombin III deficiency (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Corneal perforation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal disorder (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic graft versus host disease (Immune system disorders) | 0 (0) | 0 (0) | 2 (5)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 2 (6)
Prostate infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Evaluation (DEv) (N=3) | Phase 1: Dose Expansion (DEx) (N=10) | Phase 2: FLT3-mutated AML (N=84)
Anaemia (Blood and lymphatic system disorders) | 3 (14) | 6 (26) | 22 (107)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (7) | 9 (17) | 53 (110)
Leukopenia (Blood and lymphatic system disorders) | 2 (23) | 2 (20) | 7 (62)
Neutropenia (Blood and lymphatic system disorders) | 2 (18) | 3 (19) | 10 (65)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (27) | 2 (29) | 13 (88)
Thyroiditis chronic (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 11 (12)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 35 (50)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 5 (7) | 33 (53)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (8)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (4) | 27 (50)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 3 (4) | 25 (34)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 16 (32)
Infusion site rash (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 2 (4) | 0 (0) | 5 (5)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 6 (9)
Pain (General disorders) | 0 (0) | 0 (0) | 5 (8)
Pyrexia (General disorders) | 1 (6) | 0 (0) | 39 (66)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (2) | 0 (0) | 8 (10)
Hypogammaglobulinaemia (Immune system disorders) | 1 (2) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 17 (18)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 3 (7) | 3 (3)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4)
Device related infection (Infections and infestations) | 1 (2) | 1 (2) | 5 (5)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 4 (6)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 9 (9)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 5 (6)
Pneumonia (Infections and infestations) | 2 (3) | 5 (6) | 14 (16)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (4)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (4) | 13 (19)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 6 (7)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 4 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 37 (112)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 28 (81)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 6 (6)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 3 (4)
Blood creatinine increased (Investigations) | 0 (0) | 1 (2) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 3 (6) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 5 (13)
Liver function test abnormal (Investigations) | 2 (10) | 3 (13) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (10) | 5 (33)
Neutrophil count decreased (Investigations) | 1 (1) | 5 (21) | 27 (104)
Platelet count decreased (Investigations) | 1 (3) | 6 (33) | 29 (226)
White blood cell count decreased (Investigations) | 1 (1) | 7 (34) | 15 (84)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 9 (14)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 6 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 9 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 29 (70)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 7 (8)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 12 (16)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 6 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 8 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 6 (19)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 7 (7)
Headache (Nervous system disorders) | 0 (0) | 1 (3) | 18 (23)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 16 (32)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 11 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 9 (12)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 9 (9)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (9) | 15 (15)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (7) | 11 (21)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 11 (11)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 11 (15)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 7 (7)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 7 (9)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 32 (52)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 5 (9)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 10 (15)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 10 (16)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (10)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (6)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (7)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
Malaise (General disorders) | 0 (0) | 0 (0) | 6 (16)
Graft versus host disease (Immune system disorders) | 0 (0) | 0 (0) | 8 (9)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 5 (6)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 8 (9)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 5 (5)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2021-08-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT02310321/Prot_002.pdf
  • Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT02310321/SAP_003.pdf